CLINICAL TRIAL: NCT05582798
Title: A Proof of Concept Trial of Alpha-1 Antitrypsin Augmentation Therapy in Patients With Bronchiectasis
Brief Title: Bronchiectasis Alpha-1 Augmentation Trial- Modulating Airway Neutrophil Function
Acronym: BATMAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, James Chalmers, Professor, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.002.21
Record Dates: First submitted 2022-06-29; First posted 2022-10-17 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Bronchiectasis Adult
MeSH Terms: interventions — alpha 1-Antitrypsin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Alpha1-Proteinase Inhibitor 180mg/kg (Active Comparator): Alpha1-Proteinase Inhibitor 180mg/kg, intravenous infusion, 50mg/ml
  Interventions: Drug: Alpha 1-Proteinase Inhibitor 180mg/kg
- Alpha1-Proteinase Inhibitor 120mg/kg (Active Comparator): Alpha1-Proteinase Inhibitor 180mg/kg, intravenous infusion, 50mg/ml
  Interventions: Drug: Alpha 1-Proteinase Inhibitor 120mg/kg
- Placebo 1 (Placebo Comparator): Sodium chloride 0.9% volume to match that of Alpha1-Proteinase Inhibitor 180mg/kg, intravenous infusion.
  Interventions: Drug: Sodium chloride
- Placebo 2 (Placebo Comparator): Sodium chloride 0.9% volume to match that of Alpha1-Proteinase Inhibitor 120mg/kg, intravenous infusion.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Alpha 1-Proteinase Inhibitor 180mg/kg — alpha1-proteinase inhibitor (human) intravenous infusion
  Other Names: Prolastin-C Liquid
  Arms: Alpha1-Proteinase Inhibitor 180mg/kg
Drug: Alpha 1-Proteinase Inhibitor 120mg/kg — alpha1-proteinase inhibitor (human) intravenous infusion
  Other Names: Prolastin-C Liquid
  Arms: Alpha1-Proteinase Inhibitor 120mg/kg
Drug: Sodium chloride — Sodium chloride 09.% intravenous infusion
  Arms: Placebo 1; Placebo 2

SUMMARY:
Double-blind, randomized, cross-over trial involving 20 participants with bronchiectasis.

This trial will make an important contribution to therapeutic development in bronchiectasis by determining whether alpha-1 antitrypsin (AAT) therapy results in reduced airway inflammation and improves neutrophil function.

Patients will be randomly assigned to receive Prolastin-C 120mg/kg (n=10 patients) by weekly intravenous infusions, Prolastin-C 180mg/kg (n=10 patients) by weekly intravenous infusions or placebo (0.9% saline) for a period of 4 weeks, followed by a 3-5 week washout period and a further 4 weeks during which patients will cross-over to receive the alternative therapy.

DETAILED DESCRIPTION:
Bronchiectasis is a debilitating chronic disease associated with a vicious cycle of lung inflammation, infection and failure of mucociliary clearance.

It affects up to 566/100,000 patients in Europe and the prevalence is increasing. Excess neutrophil proteinase activity is central to the pathogenesis of bronchiectasis. Neutrophil elastase is released from activated neutrophils recruited to the bronchiectasis lung and exacerbates inflammation through multiple mechanisms. These include stimulating goblet cell hyperplasia and mucus production, altering of ciliary beat frequency, preventing neutrophil phagocytosis of pathogens through cleavage of phagocytic receptors and preventing apoptotic cell clearance through the cleavage of phosphatidylserine. Neutrophil elastase activity in the bronchiectasis lung is increased because the concentration of elastase released from neutrophils exceeds the inhibitory capacity of the natural anti-proteinase defences of the lung. Of these, alpha-1 proteinase inhibitor accounts for approximately 90% of the inhibitory capacity. The adverse effects of excess proteinase activity are observed in genetic alpha-1 antitrypsin deficiency (A1ATD) where patients develop progressive emphysema, lung function decline, and bronchiectasis.

The majority of bronchiectasis patients do not have genetic A1ATD but do have functional alpha-1 antitrypsin deficiency because elastase activity exceeds the available alpha-1 antitrypsin in the lung. There are currently no licensed treatments that directly target excessive neutrophil elastase activity in bronchiectasis.

The investigators hypothesize that augmentation of alpha-1 proteinase inhibitor could have beneficial effects in patients with bronchiectasis who have elevated sputum neutrophil elastase activity. Currently, licensed alpha-1 antitrypsin augmentation therapy is given by intravenous infusions on a weekly basis to patients with genetic A1ATD. Inhaled alpha-1 proteinase inhibitor has been used previously in trials in cystic fibrosis. While inhaled alpha1 proteinase inhibitor may have a role in the future in bronchiectasis, the investigators are proposing to conduct a trial of intravenous administration as a proof-of-concept due to the known safety profile of the licensed product and due to increasing evidence that neutrophils in bronchiectasis are dysfunctional in the systematic circulation, with an activated phenotype and evidence of systematic elastin degradation measured by serum desmosine.

The investigators propose a proof-of-concept trial which will gather important data to determine the feasibility and scientific value of a future efficacy trial of alpha-1 proteinase inhibitor augmentation in bronchiectasis.

There is an urgent unmet need for new therapies in bronchiectasis, a point that has been made by physicians, patients and regulators. There are currently no licensed therapies and off-label treatments have limited effectiveness leaving a high disease burden. European registry data shows that approximately 50% of patients experience two or more exacerbations per year and 1/3 experience at least one admission to hospital for severe exacerbations each year. Patients with elevated neutrophil elastase activity in sputum experience more rapid decline in lung function, more exacerbations and worse quality of life, yet there are no treatments which directly target lung inflammation in bronchiectasis.

This trial will make an important contribution to therapeutic development in bronchiectasis by determining whether alpha-1 antitrypsin (AAT) therapy results in reduced airway inflammation and improves neutrophil function. This in turn will inform future therapeutic development in bronchiectasis including determining the potential for a future definitive efficacy and safety trial in bronchiectasis patients. This is the "treatable trait" that the investigators aim to target with AAT administration and this approach of treatment guided by a point-of-care biomarker will be a further innovative aspect of the trial.

This is a double-blind, randomized, cross-over trial involving 20 participants with bronchiectasis. The trial will consist of a screening period of up to 35 days followed by a total trial duration of up to 13 weeks. Patients will be randomly assigned to receive Prolastin-C 120mg/kg (n=10 patients) by weekly intravenous infusions, Prolastin-C 180mg/kg (n=10 patients) by weekly intravenous infusions or placebo (0.9% saline) for a period of 4 weeks, followed by a 3-5 week washout period and a further 4 weeks during which patients will cross-over to receive the alternative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Bronchiectasis on high resolution computerised tomography (CT) scan affecting 1 or more lobes
* Sputum neutrophil elastase activity greater than or equal to 7 µg/ml on neutrophil elastase assay at the screening visit*
* Daily sputum production as determined by the researcher from the patient's self-report
* Able to provide a sputum sample at the screening and randomization visits either spontaneously
* Ability to give informed consent
* Able to perform all trial procedures with minimal assistance
* Willing to have pregnancy testing, if appropriate

Exclusion Criteria:

* Severe alpha-1 antitrypsin deficiency (<57 mg/dl in serum) regardless of genotype#
* Immunoglobulin A (IgA) deficient patients with antibodies against IgA
* History of anaphylaxis or other severe systemic reaction to Alpha1-Proteinase Inhibitor
* Primary diagnosis of Chronic Obstructive Pulmonary Disease (COPD) in the opinion of the investigator
* Primary Diagnosis of asthma in the opinion of the investigator
* Active allergic bronchopulmonary aspergillosis, NTM, immunodeficiency or another aetiology of bronchiectasis requiring a specific treatment
* Treatment with antibiotic therapy for an exacerbation of bronchiectasis (other than long term oral or inhaled antibiotics at stable dose) in the 4 weeks prior to randomization
* Cystic fibrosis
* Unstable cardiac disease in the opinion of the investigator
* Congestive cardiac failure and in the opinion of the investigator should not receive iv infusions.
* Traction bronchiectasis due to interstitial lung disease
* Current smoker
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of intravenous alpha-1 proteinase inhibitor on sputum neutrophil elastase activity | Baseline and 4 weeks
  Change from baseline in sputum neutrophil elastase activity measured in units/ml

SECONDARY OUTCOMES:
To determine the effect of intravenous alpha-1 proteinase inhibitor on neutrophil function | Baseline and 4 weeks
  Change from baseline in alpha-1 antitrypsin levels by immunoassay
To determine the effect of intravenous alpha-1 proteinase inhibitor on neutrophil function | Baseline and 4 weeks
  Sputum neutrophil extracellular traps measured using immunoassay
To determine the effect of intravenous alpha-1 proteinase inhibitor on neutrophil function | Baseline and 4 weeks
  Activity of cathepsin G and proteinase-3 in sputum
To determine the effect of intravenous alpha-1 proteinase inhibitor on neutrophil function | Baseline and 4 weeks
  Sputum neutrophil cell counts
To determine the effect of intravenous alpha-1 proteinase inhibitor on neutrophil function | Baseline and 4 weeks
  Sputum neutrophil migration
To determine the effect of intravenous alpha-1 proteinase inhibitor on neutrophil function | Baseline and 4 weeks
  Sputum neutrophil degranulation
To determine the effect of intravenous alpha-1 proteinase inhibitor on neutrophil function | Baseline and 4 weeks
  Sputum neutrophil phagocytosis
To determine clinical benefits of alpha-1 proteinase inhibitor | Baseline and 4 weeks
  Spirometry: forced expiratory volume in 1 minute (FEV1)
To determine clinical benefits of alpha-1 proteinase inhibitor | Baseline and 4 weeks
  Spirometry: forced vital capacity (FVC)
To determine clinical benefits of alpha-1 proteinase inhibitor | Baseline and 4 weeks
  Spirometry: forced expiratory flow 25-75% (FEV25-75)
To determine clinical benefits of alpha-1 proteinase inhibitor | Baseline and 4 weeks
  Spirometry: forced expiratory volume in 1 minute/forced vital capacity (FEV1/FVC)
To determine clinical benefits of alpha-1 proteinase inhibitor | Baseline and 4 weeks
  Spirometry: forced expiratory volume in 1 minute (FEV1); forced vital capacity (FVC); forced expiratory flow 25-75% (FEV25-75); forced expiratory volume in 1 minute/forced vital capacity (FEV1/FVC)
To determine safety and tolerability of intravenous alpha-1 proteinase inhibitor administration | 4 weeks
  Adverse events, serious adverse events and trial treatment withdrawals will be recorded and a comparison made between the 4 treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: James Chalmers, Principal Investigator — University of Dundee
Locations (1):
- NHS Tayside, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No